CLINICAL TRIAL: NCT04120350
Title: R2-MTX Regimen Combined With Lenalidomide Maintenance as Frontline Therapy for Primary Central Nervous System Lymphoma: a Multicenter Prospective Single Arm Trial.
Brief Title: R2-MTX With Lenalidomide Maintenance in Newly-diagnosed PCNSL：a Multicenter Phase Ib/II Stuty
Acronym: REMLA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Xuanwu Hospital, Beijing (Other); Peking University Third Hospital (Other); Beijing Hospital (Other Government); Peking University First Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-004
Record Dates: First submitted 2019-09-28; First posted 2019-10-09 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: lenalidomide; rituximab; methorexate; Primary Central Nervous System Lymphoma; maintenance therapy
MeSH Terms: interventions — Methotrexate; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R2-MTX-LEN (Experimental): Phase Ib：Experimental arm will be treated with R2-MTX regimen for 6 cycles as initiate induction, the dose of lenalidomide was escalated from 15mg， 20mg， 25mg to test DLT by 3+3 design, meanwhile the dose of rituximab and methotrexate is fixed. If the patients achieved CR or PR by MRI and CSF evaluation, they processed to lenalidomide maintenance for 2 years.
  Phase II: the patients will be treated by fixed dose of R2-MTX regimen (established lenalidomide dose from phase Ib study) for 6 cycles. the efficiency evaluation will be performed every 2 cycles, the patients who achieved CR or PR will finish the total 6 cycles of induction therapy, then begin the stage of lenalidomide maintenance for 2 years. Follow-ups should be taken for 5 years.
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Methotrexate — 3.5g/m2 intravenous infusion for 4 hours in d1, every 21 days for 1 cycle. 6 cycles will be prescribed as protocol
Drug: Rituximab — 375mg/m2 intravenous infusion d1, every 21 days for 1 cycle. 6 cycles will be prescribed as protocol
Drug: Lenalidomide — In phase 1b study, a 3+3 design dose- escalation will be taken. 3 levels should be tested, 15/20/25mg orally d1-14, every 21 days for 1 cycle. 6 cycles will be prescribed as protocol.
  [update 02-Jun-2020: the phase Ib trial has finished,and no MDT was obsevered in 25mg group. So the recommanded phase II dose was 25mg.] In phase II study, 25mg daily is considered as an experiment dose for the induction cycles.
  In both phase Ib and II study, the does of lenalidomide maintenance is fixed to 25mg orally d1-21 every 28 days for 1 cycle. The duration of maintenance is 2 years.

SUMMARY:
This is a multicenter prospective single arm phase Ib/II study, and the purpose of this study is to evaluate the safety and efficiency of R2-MTX regimen (rituximab & lenalidomide & methotrexate) combined with lenalidomide maintenance in newly-diagnosed primary central nervous system lymphoma. 2-year Progression free survival (PFS) of the cohort is the primary endpoint.

DETAILED DESCRIPTION:
There are 2 section of this trial. Step1 is a phase Ib study.The patients will be treated with R2-MTX regimen （Rituximab 375mg/m2 IV d0, methotrexate 3.5g/m2 civ d1, lenalidomide 15-25mg d1-14, 21 days per cycle) as induction regimen.The dose of rituximab and methotrexate is fixed dose. This is a 3+3 design Ib phase dose-escalation study to determined the maximum tolerated dose(MTD) of lenalidomide dose in combined regimen. 3 levels of lenalidomide dose will be investigated, 15mg, 20mg and 25mg. If the DLT is not found, the dose of 25mg qd will be used for phase II trial.

[update 02-Jun-2020：the recommended phase II doses is 25mg d1-14]

Step 2 is a single-arm phase 2 study with fixed does of R2-MTX regimen in newly-diagnosed PCNSL patients. The response will be evaluated every 2 cycles. Patients who achieved complete remission (CR) or partial remission (PR) will receive further treatment, and there are 6 cycles of R2-MTX regimen for the induction. The patients with stable disease (SD) or progressed disease (PD) will withdraw from the trial and receive salvage regimens. After total 6 induction cycles, the investigators evaluate the efficiency again, the patients with CR or PR will go to lenalidomide maintenance for 2 years or until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion. And the patients with SD or PD will receive salvage regimen.

[update 02-Jun-2020：Younger patients(≤60 years) who achieve PR after 6 cycles of induction therapy will be candidates of high-dose chemotherapy and stem cell rescue. Lenalidomide maintenance will be administed after the high-dose chemotherapy. Older patients(>60 years) who achieve PR after 6 cycles of induction will go to lenalidomide maintenance directly.] During following-up, surveillance examination and brain magnetic resonance imaging (MRI) scans can be performed every 3 months up to the first 2 years, followed by doctor visit every 6 months up to 5 years or the disease relapses.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed primary vitreoretinal lymphoma
* ECOG≤2
* creatinine clearance rate (CCR) ≥ 50ml/h, according to Cockcroft-Gault
* Total bilirubin < 2 upper limits of normal, alanine aminotransferase（ALT） < 3 upper limits of normal
* HIV-Ab negative
* Sign the Informed consent
* Women of childbearing potential must understand that the study medication could have a potential teratogenic risk. They should undergo complete contraception during the study period.
* Male subjects must agree to use condoms throughout study drug therapy.

Exclusion Criteria:

* Pre-existing uncontrolled active infection
* Clinical evidence of grade 3 or 4 heart failure as defined by the New York Heart Association criteria
* systemic lymphoma involved CNS
* Pregnancy or active lactation
* Co-existing tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
2 years progression-free survival | From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow-up without relapsing

SECONDARY OUTCOMES:
2 years overall survival | From date of signing the informed consent until the date of death from any cause, whichever came first, assessed up to 2 years
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow-up alive
dose-limiting toxicity（DLT） | from the start of the first dose of lenalidomide to the finish of first cycle of induction(21 days for each cycle).
  all treatment-related, critically relevant grade 3/4 adverse event (AE) that occured in the first 21 days after the start of the first treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Daobin Zhou, Beijing, Dongcheng District, China

IPD SHARING:
Plan to Share IPD: No